CLINICAL TRIAL: NCT00988468
Title: Effects of Manual Therapy Versus Therapeutic Exercise on Knee Osteoarthritis: A Randomized Control Trial
Brief Title: Manual Therapy Versus Exercise on Knee Osteoarthritis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study failed to recruit a sufficient number of subjects in the time anticipated.
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Daniel R. Poulsen, II/Assistant Professor, Texas Tech University Health Sciences Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: L10-004
Record Dates: First submitted 2009-09-30; First posted 2009-10-02 (Estimated); Last update posted 2010-11-16 (Estimated); Status verified 2010-11

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Manual Therapy; Therapeutic Exercise; Ultrasound; Effusion
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Musculoskeletal Manipulations; Exercise Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Manual Therapy (Experimental): Subjects will receive oscillatory (grade 1 & 2) manual knee mobilization for 15 minutes at various knee range of motion positions.
  Interventions: Procedure: Manual Therapy
- Therapeutic Exercise (Experimental): Subjects will perform 15 minutes of combined resistance exercise and aerobic exercise.
  Interventions: Behavioral: Therapeutic Exercise
- Control (Placebo Comparator): Subjects will watch a 15 minute instructional video on a health topic.
  Interventions: Behavioral: Video Observation

INTERVENTIONS:
Procedure: Manual Therapy — Grade 1 and 2 oscillatory manual mobilization of the tibiofemoral joint at various ranges of motion.
  Arms: Manual Therapy
Behavioral: Therapeutic Exercise — Subjects will perform 5 minutes of lower extremity cycle ergometer with minimal resistance followed by 10 minutes of resistance exercise to the quadriceps at 3 tibiofemoral positions (0 degrees, 30 degrees and 60 degrees of knee flexion).
  Arms: Therapeutic Exercise
Behavioral: Video Observation — Subjects will watch a 15 minute video on a health topic unrelated to knee osteoarthritis.
  Arms: Control

SUMMARY:
Earlier research has shown that exercising while receiving manual therapy improves function and reduces pain in people with knee osteoarthritis. However, very little is known about the mechanisms by which manual therapy and exercise reduce pain and improve function. This study will ask subjects with knee osteoarthritis to receive one of the following interventions: (1) no treatment, (2) exercise only, or (3) manual therapy only. Measures will be taken of the patient's knee range of motion, knee swelling and pain before and after receiving the intervention. These measures will be analyzed to determine what effect exercise and manual therapy applied to the knee have on improving knee range of motion and reducing knee pain and swelling. Swelling will be measured using an ultrasound device which is used to take pictures inside the knee. This type of ultrasound measurement is painless and harmless.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of knee osteoarthritis.

Exclusion Criteria:

* Inability to ambulate at least 100 feet, ride a stationary bicycle for at least 10 minutes, or lie in the prone position for at least 10 minutes,
* Intra-articular knee injection within one month of study inception,
* A history of exercise induced or uncontrolled angina within three months of the study entry,
* Severe dyspnea at rest,
* Previous bilateral total knee arthroplasty,
* Pregnancy, OR
* The absence of knee pain at the time of recruitment for the study.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-10; Primary Completion 2010-05 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Suprapatellar effusion measured via diagnostic ultrasound | Outcome measure will be measured 1 minute prior to intervention and 1 minute after intervention.

SECONDARY OUTCOMES:
Pain Visual Analog Scale | Outcome measure will be measured 3 minutes prior to intervention and 3 minutes after intervention.
Goniometric knee arc range of motion | Outcome measure will be measured 5 minutes prior to intervention and 5 minutes after intervention.
Western Ontario and McMaster Universities Index of osteoarthritis of the knee | Outcome measure will be measured 12 minutes prior to intervention and 7 minutes after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Poulsen, PhD, Principal Investigator — Texas Tech University Health Sciences Center
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, Texas, United States

REFERENCES:
- [Background] Lawrence RC, Felson DT, Helmick CG, Arnold LM, Choi H, Deyo RA, Gabriel S, Hirsch R, Hochberg MC, Hunder GG, Jordan JM, Katz JN, Kremers HM, Wolfe F; National Arthritis Data Workgroup. Estimates of the prevalence of arthritis and other rheumatic conditions in the United States. Part II. Arthritis Rheum. 2008 Jan;58(1):26-35. doi: 10.1002/art.23176. PMID 18163497
- [Background] Zhang W, Moskowitz RW, Nuki G, Abramson S, Altman RD, Arden N, Bierma-Zeinstra S, Brandt KD, Croft P, Doherty M, Dougados M, Hochberg M, Hunter DJ, Kwoh K, Lohmander LS, Tugwell P. OARSI recommendations for the management of hip and knee osteoarthritis, Part II: OARSI evidence-based, expert consensus guidelines. Osteoarthritis Cartilage. 2008 Feb;16(2):137-62. doi: 10.1016/j.joca.2007.12.013. PMID 18279766
- [Background] Hunter DJ, Felson DT. Osteoarthritis. BMJ. 2006 Mar 18;332(7542):639-42. doi: 10.1136/bmj.332.7542.639. No abstract available. PMID 16543327
- [Background] Ottawa panel evidence-based clinical practice guidelines for therapeutic exercises and manual therapy in the management of osteoarthritis. Phys Ther. 2005 Sep;85(9):907-71. PMID 16117601
- [Background] Hoeksma HL, Dekker J, Ronday HK, Heering A, van der Lubbe N, Vel C, Breedveld FC, van den Ende CH. Comparison of manual therapy and exercise therapy in osteoarthritis of the hip: a randomized clinical trial. Arthritis Rheum. 2004 Oct 15;51(5):722-9. doi: 10.1002/art.20685. PMID 15478147
- [Background] Moss P, Sluka K, Wright A. The initial effects of knee joint mobilization on osteoarthritic hyperalgesia. Man Ther. 2007 May;12(2):109-18. doi: 10.1016/j.math.2006.02.009. Epub 2006 Jun 13. PMID 16777467
- [Background] Wright A. Hypoalgesia post-manipulative therapy: a review of a potential neurophysiological mechanism. Man Ther. 1995 Nov;1(1):11-6. doi: 10.1054/math.1995.0244. PMID 11327789
- [Background] Sambajon VV, Cillo JE Jr, Gassner RJ, Buckley MJ. The effects of mechanical strain on synovial fibroblasts. J Oral Maxillofac Surg. 2003 Jun;61(6):707-12. doi: 10.1053/joms.2003.50141. PMID 12796883
- [Background] Knott EM, Tune JD, Stoll ST, Downey HF. Increased lymphatic flow in the thoracic duct during manipulative intervention. J Am Osteopath Assoc. 2005 Oct;105(10):447-56. PMID 16314677
- [Background] Coates G, O'Brodovich H, Goeree G. Hindlimb and lung lymph flows during prolonged exercise. J Appl Physiol (1985). 1993 Aug;75(2):633-8. doi: 10.1152/jappl.1993.75.2.633. PMID 8226462
- [Background] Havas E, Lehtonen M, Vuorela J, Parviainen T, Vihko V. Albumin clearance from human skeletal muscle during prolonged steady-state running. Exp Physiol. 2000 Nov;85(6):863-8. PMID 11187981
- [Background] de Miguel Mendieta E, Cobo Ibanez T, Uson Jaeger J, Bonilla Hernan G, Martin Mola E. Clinical and ultrasonographic findings related to knee pain in osteoarthritis. Osteoarthritis Cartilage. 2006 Jun;14(6):540-4. doi: 10.1016/j.joca.2005.12.012. PMID 16735196
- [Background] Conaghan P, D'Agostino MA, Ravaud P, Baron G, Le Bars M, Grassi W, Martin-Mola E, Wakefield R, Brasseur JL, So A, Backhaus M, Malaise M, Burmester G, Schmidely N, Emery P, Dougados M. EULAR report on the use of ultrasonography in painful knee osteoarthritis. Part 2: exploring decision rules for clinical utility. Ann Rheum Dis. 2005 Dec;64(12):1710-4. doi: 10.1136/ard.2005.038026. Epub 2005 May 5. PMID 15878902
- [Background] Altman R, Asch E, Bloch D, Bole G, Borenstein D, Brandt K, Christy W, Cooke TD, Greenwald R, Hochberg M, et al. Development of criteria for the classification and reporting of osteoarthritis. Classification of osteoarthritis of the knee. Diagnostic and Therapeutic Criteria Committee of the American Rheumatism Association. Arthritis Rheum. 1986 Aug;29(8):1039-49. doi: 10.1002/art.1780290816. PMID 3741515
- [Background] Dexter F, Chestnut DH. Analysis of statistical tests to compare visual analog scale measurements among groups. Anesthesiology. 1995 Apr;82(4):896-902. doi: 10.1097/00000542-199504000-00012. PMID 7717561
- [Background] Duncan GH, Bushnell MC, Talbot JD, Evans AC, Meyer E, Marrett S. Pain and activation in the thalamus. Trends Neurosci. 1992 Jul;15(7):252-3. doi: 10.1016/0166-2236(92)90062-d. No abstract available. PMID 1381119
- [Background] Duncan GH, Bushnell CM, Lavigne GJ. Comparison of verbal and visual analogue scales for measuring the intensity and unpleasantness of experimental pain. Pain. 1989 Jun;37(3):295-303. doi: 10.1016/0304-3959(89)90194-2. PMID 2755711
- [Background] Jan MH, Chai HM, Wang CL, Lin YF, Tsai LY. Effects of repetitive shortwave diathermy for reducing synovitis in patients with knee osteoarthritis: an ultrasonographic study. Phys Ther. 2006 Feb;86(2):236-44. PMID 16445337
- [Background] Deyle GD, Allison SC, Matekel RL, Ryder MG, Stang JM, Gohdes DD, Hutton JP, Henderson NE, Garber MB. Physical therapy treatment effectiveness for osteoarthritis of the knee: a randomized comparison of supervised clinical exercise and manual therapy procedures versus a home exercise program. Phys Ther. 2005 Dec;85(12):1301-17. PMID 16305269
- [Background] Miyaguchi M, Kobayashi A, Kadoya Y, Ohashi H, Yamano Y, Takaoka K. Biochemical change in joint fluid after isometric quadriceps exercise for patients with osteoarthritis of the knee. Osteoarthritis Cartilage. 2003 Apr;11(4):252-9. doi: 10.1016/s1063-4584(02)00372-2. PMID 12681951